CLINICAL TRIAL: NCT06153797
Title: Randomized Controlled Trial of a Positive Psychology Based Intervention (PATH-C) for Caregivers of Hematopoietic Stem Cell Transplant Survivors
Brief Title: A Positive Psychology Based Intervention (PATH-C) for Caregivers of HSCT Survivors
Acronym: PATH-C
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Robert Wood Johnson Foundation (Other); American Society of Hematology (Other)
Responsible Party: Principal Investigator, Hermioni L.Amonoo, MD, MPP, MPH, Director, Well-Being and Cancer Research Program, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-509
Record Dates: First submitted 2023-11-23; First posted 2023-12-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hematologic Malignancy; Caregiver
Keywords: Hematologic Malignancy; Hematopoietic Stem Cell Transplant; Caregivers of Patients with Cancer; Positive Psychology Intervention
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is a single-site randomized efficacy trial of the PATH-C intervention in 80 caregivers of patients with hematologic malignancies undergoing hematopoietic stem cell transplantation. Participants will be recruited from the Dana-Farber Cancer Institute and randomized in a 1:1 fashion, stratified by transplant type (autologous versus allogeneic), to assign each participant to either PATH-C versus usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PATH-C (Experimental): Participants will be recruited from the Dana-Farber Cancer Institute and randomized in a 1:1 fashion, stratified by transplant type (autologous versus allogeneic), to PATH-C versus usual care.
  Caregivers of patients undergoing HSCT will receive the PATH-C intervention to learn to reflect on their positive emotions and consistently use and incorporate positive psychology exercises in their daily routine, as well as learn how to set goals and track their physical activity (i.e., with an activity tracker) daily while caring for a loved one undergoing HSCT.
  Participants will complete questionnaires (in person, over the computer or telephone, or by mail) at predetermined days per protocol.
  Interventions: Behavioral: PATH-C
- Usual Care (No Intervention): Participants will be recruited from the Dana-Farber Cancer Institute and randomized in a 1:1 fashion, stratified by transplant type (autologous versus allogeneic), to PATH-C versus usual care.
  Participants will complete questionnaires (in person, over the computer or telephone, or by mail) at predetermined days per protocol.
  Participants in the usual care arm will receive their usual support from the HSCT team as caregivers of patients undergoing HSCT, including all routine supportive care resources (e.g., support from social work) offered by the HSCT team.
  Patients in the usual care and PATH-C groups will be permitted to use all supportive care services per standard care. The investigators will track referrals to supportive care services in both groups by reviewing the Electronic Health Record (EHR).

INTERVENTIONS:
Behavioral: PATH-C — PATH-C, a phone-delivered positive psychology intervention for caregivers of patients undergoing HSCT, consists of the following nine sessions: 1) Enhancing gratitude and increasing awareness for physical activity; 2) Expressing gratitude and goal setting for physical activity; 3) Integrating gratitude and goals for physical activity; 4) Personal strengths and environmental scan to enhance physical activity; 5) Enhancing strengths via reflection on past successes; 6) Integrating strengths to enhance well-being and physical activity; 7) Engaging in enjoyable and meaningful activities; 8) Promoting optimism and integrating long-term activity habits; 9) Integrating meaning for sustainable physical activity goals. Each session takes about 30 minutes, and a trained interventionist will guide participants to complete the sessions.
  Arms: PATH-C

SUMMARY:
The goal of this randomized clinical trial is to evaluate whether a positive psychology intervention (PATH-C) can improve psychological well-being, quality of life, and physical activity in caregivers of patients undergoing hematopoietic stem cell transplantation (HSCT).

DETAILED DESCRIPTION:
Family and friend caregivers are vital care providers throughout the entire care continuum for patients with hematologic malignancies undergoing hematopoietic stem cell transplantation (HSCT). These caregivers must manage multiple time-consuming responsibilities, including monitoring vital signs and side effects of treatment, administering medications, and coordinating transportation to and from medical appointments. The substantial caregiving burden among caregivers of patients undergoing HSCT is associated with increased symptoms of depression, anxiety, and fatigue. Symptoms such as fatigue and depression in HSCT caregivers may undermine attempts to maintain regular physical activity routines, which may impact essential health outcomes such as cardiovascular health.

With persistent shortages in the mental health workforce needed to address these psychological needs of HSCT caregivers adequately, remotely-delivered psychosocial interventions offer an innovative approach to overcome the unmet psychological needs of this population. Hence, the investigators developed a remotely-delivered positive psychology intervention, Positive Affect in the Transplantation of Hematopoietic Stem Cells for Caregivers (PATH-C), tailored to the unique psychological needs of HSCT caregivers. With this study, the investigators will establish the impact of PATH-C on participant-reported outcomes compared to usual care.

The study will use validated questionnaires to measure caregivers' quality of life, caregiver burden, psychological distress symptoms, positive psychological well-being (e.g., positive affect, gratitude), and self-management targets (e.g., coping, self-efficacy). The study will also use the validated ActiGraph GT3X+ accelerometer to measure minutes/day of moderate-to-vigorous physical activity, light activity, and sedentary leisure time.

ELIGIBILITY:
Inclusion Criteria:

* Adult caregivers (aged 18 years and older) of patients undergoing allogeneic or autologous HSCT at Dana-Farber Cancer Institute for a hematologic malignancy.
* A relative or a friend who either lives with the patient or has in-person contact with them at least twice per week and is identified as the primary caregiver for HSCT.
* Ability to speak English and able to complete questionnaires with minimal assistance of an interpreter as this is a feasibility trial of the PATH-C intervention which is currently only available in English.

Exclusion Criteria:

* Caregivers of patients undergoing HSCT for benign hematologic conditions.
* Caregivers with acute or unstable psychiatric conditions which the treating transplant clinician believes prohibits informed consent or compliance with study procedures.
* Cognitive deficits impeding a caregiver's ability to provide informed consent or participate adequately in the study assessed via a commonly used 6-item cognitive assessment with the Brief Interview for Mental Status (BIMS) screening tool that is sensitive and specific for screening for cognitive impairment in research participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
PATH-C Intervention Feasibility | Up to 10 weeks
  PATH-C Intervention Feasibility is defined as >60% of eligible participants enrolling in the study and >60% of enrolled participants who start the intervention completing at least 6/9 intervention sessions.

SECONDARY OUTCOMES:
PATH-C Intervention Acceptability | Up to 10 weeks
  Acceptability will be measured using weekly ratings of the ease and utility of each exercise (0=very difficult/not helpful; 10=very easy/very helpful) and will use a threshold of a mean combined score of 7.0/10.0.
Physical activity longitudinally based on ActiGraph GT3X+ accelerometer | Up to 20 weeks (+/- 28 days)
  Compare physical activity levels using the ActiGraph GT3X+ accelerometer between the two groups.
  Greater steps/day and lower sedentary leisure time indicate greater physical activity.
Caregiver Quality of Life based on the CarGOQOL | Up to 20 weeks (+/- 28 days)
  Compare caregiver quality of life using the 29-item CareGiver Oncology Quality of Life questionnaire (CarGOQOL) between the two groups.
  Higher scores on the CarGOQOL (normalized score range, 1-100) indicate better quality of life.
Anxiety Symptoms based on the HADS-Anxiety Subscale | Up to 20 weeks (+/- 28 days)
  Compare anxiety symptoms using the 7-item Hospital Anxiety and Depression Scale-Anxiety (HADS-A) subscale between the two groups.
  The HADS-A subscale ranges from 0-21, with higher scores indicating worse anxiety symptoms.
Depression Symptoms based on the HADS-Depression Subscale | Up to 20 weeks (+/- 28 days)
  Compare depression symptoms using the 7-item Hospital Anxiety and Depression Scale-Depression (HADS-D) subscale between the two groups.
  The HADS-D subscale ranges from 0-21, with higher scores indicating worse depression symptoms.
Caregiving Burden based not the Caregiver Reaction Assessment (CRA) | Up to 20 weeks (+/- 28 days)
  Compare caregiving burden using the 24-item Caregiver Reaction Assessment (CRA) between the two groups.
  The CRA ranges from 24 to 120, with higher scores indicating greater caregiving burden.

OTHER OUTCOMES:
Optimism | Up to 20 weeks (+/- 28 days)
  Compare optimism using the 10-item Life Orientation Test-Revised (LOT-R) between the two groups.
  The LOT-R ranges from 0 to 24, with higher scores indicating greater optimism.
Positive Affect | Up to 20 weeks (+/- 28 days)
  Compare positive affect using the 15-item Patient-Reported Outcomes Measurement Information System (PROMIS) Positive Affect Short Form between the two groups.
  The PROMIS Positive Affect Short Form ranges from 15 to 75, with higher scores indicating greater positive affect.
Life Satisfaction | Up to 20 weeks (+/- 28 days)
  Compare life satisfaction using the 10-item Patient-Reported Outcomes Measurement Information System (PROMIS) General Life Satisfaction Questionnaire between the two groups.
  The PROMIS General Life Satisfaction Questionnaire ranges from 10 to 60, with higher scores indicating greater satisfaction with life.
Gratitude | Up to 20 weeks (+/- 28 days)
  Compare gratitude using the 6-item Gratitude Questionnaire between the two groups.
  The Gratitude Questionnaire ranges from 6 to 42, with higher scores indicating a stronger propensity for experiencing gratitude in daily life.
Flourishing | Up to 20 weeks (+/- 28 days)
  Compare flourishing using the 8-item Flourishing Scale between the two groups.
  The Flourishing Scale ranges from 8 to 56, with higher scores indicating having more psychological resources and strengths.
Self-Efficacy | Up to 20 weeks (+/- 28 days)
  Compare self-efficacy using the Cancer Self-Efficacy Scale-transplant (CASE-t) between the two groups.
  The CASE-t ranges from 0 to 170, with higher scores indicating greater self-efficacy.
Perceived Coping Skills | Up to 20 weeks (+/- 28 days)
  Compare coping skills using the Measure of Current Status (MOCS-A) between the two groups.
  The MOCS-A ranges from 0 to 52, with higher scores indicating having more coping skills.
Stress Resilience | Up to 20 weeks (+/- 28 days)
  Compare stress resilience using the 6-item Brief Resilience Scale (BRS) between the two groups.
  The BRS ranges from 6 to 30, with higher scores indicating greater stress resilience.
Locus of Control | Up to 20 weeks (+/- 28 days)
  Compare locus of control using the Multidimensional Health Locus of Control (MHLC) scale, Form A between the two groups.
  The MHLC Form A ranges from 6 to 36 for each locus of control category (internal, powerful others, or chance), and higher scores suggest greater belief in each category as the source of health locus of control.

CONTACTS AND LOCATIONS:
Overall Officials: Hermioni Amonoo, MD, MPP, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber/Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to the Sponsor, Investigator, or designee. The protocol and statistical analysis plan will be made available on ClinicalTrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the study investigator at hermioni_amonoo@dfci.harvard.edu